CLINICAL TRIAL: NCT02060136
Title: Validation of Electronic Recording of Lower Urinary Tract Symptoms (LUTS) in Men
Brief Title: Electronic Method for Recording Lower Urinary Tract Symptoms
Status: Completed | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Principal Investigator, Vaclav Prochazka, MD, PhD. MSc, Chief research officer, University Hospital Ostrava
Other Study IDs: SUF LUTS
Record Dates: First submitted 2014-01-27; First posted 2014-02-11 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: Electronic micturition chart, validation
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study group: Men presenting to the urology clinic with lower urinary tract symptoms

SUMMARY:
Urinary diaries have proven to be beneficial in assessing lower urinary tract symptoms (LUTS), however they have not achieved widespread acceptance. The likely reason is the fact that the pen and paper diaries are labor intensive for both patient (need to carry a pen and paper and record each event) and doctor (need to transfer, summarize and analyze the data).

Hypothesis: Electronic voiding diary, would automate the recording and analysis of data, expedite the process, improve its accuracy and cost effectiveness.

Electronic recording of lower urinary tract symptoms (SUF) uses wireless phone and web based technologies to record LUTS remotely and store the data on a secure website which can be accessed by the doctor or patient whenever needed. The goal of this study was to compare its validity and reliability to the traditional micturition chart (MC) recording method - the current gold standard where the patient records the time of micturition and degree of urgency using a pen and paper.

DETAILED DESCRIPTION:
SUF records the sound of the urine stream striking the water in a toilet bowl. This generates a sound file, which resembles the standard uroflowmetry recording. The degree of urgency is recorded by pressing the number 1-5 on the key pad which corresponds to the 5-point urgency scale. Urgency is recorded immediately following micturition or whenever experiencing urgency without bladder emptying. A dedicated server runs a program, which automatically processes incoming data. All data recorded from an individual is stored prospectively, in separate files, on a secure website. Each record is associated with a time stamp, providing information on urinary frequency.

A pen and pencil MC will be used to record baseline parameters (voiding urgency and frequency). Quality of life (QoL) will be evaluated using International Prostate Symptom Score (IPSS) Questionnaire, and two standardized questions: Quality of Life due to Urinary Symptoms (QoL US) and Patient Perception of Bladder Condition (PPBC).

Time frame: Participants were followed for the duration of the study which consists of two three day periods when every micturition event and lower urinary tract symptom not associated with micturition was recorded. An expected average time will be 6 days.

Twenty nine men, average age 67.8 years (range 49 - 80), which presented to the urology clinic with LUTS, were included in the study. After signing the informed consent, patients will be asked to record every micturition and degree of urgency using SUF for a period of 3 days. They will then be asked to record their frequency of micturition and the degree of every episode of urgency using a pen and paper MC for an equal length of time. The efficacy of recording LUTS with each method will be analyzed and compared. The content validity of SUF (assessment of whether the instrument makes sense to patients), will be assessed at the conclusion of the study when all patients will be interviewed one-on-one by a specialized research nurse. Patients will be asked to state their preference for one of the two diaries, and disclose the number of events they forgot to or could not record. The construct validity (relationship between the recorded data and underlying theories) will be evaluated by the correlation of symptoms recorded with SUF or MC based on QoL measures. The results of this study will be compared to previously published evidence, suggesting that more severe LUTS are associated with a lower score on the health related QoL questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Men seeking treatment for lower urinary tract symptoms

Exclusion Criteria:

* none

Ages: 45 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men presenting to the urology clinic with lower urinary tract symptoms
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2013-06; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the level of accuracy and adherence to the study protocol | January - February 2014 (1 month)
  Asses a difference between average number of micturition events, frequency, and degree of urgency episodes recorded using SUF and MC, to determine is SUF provides equally relevant information to that obtained by the standard approach.
  User compliance will be assessed though recording the number of patients who forgot to record micturitions and urgency episodes using SUF versus MC.

SECONDARY OUTCOMES:
User preference | January - February (1 month)
  The content validity of SUF (assessment of whether the instrument makes sense to patients), will be assessed at the conclusion of the study when all patients will be interviewed one-on-one by a specialized research nurse. Patients will be asked to state their preference for one of the two diaries.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Krhut, MD, PhD, Principal Investigator — Ostrava University
Locations (1):
- Department of Urology, Ostrava, Nothern Moravia, Czechia